CLINICAL TRIAL: NCT07206888
Title: Advanced Ultrasound Beamforming Methods for Breast Imaging
Brief Title: Advanced Ultrasound Signal Processing of Suspicious Breast Images
Acronym: AUSPICIOUS
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00127110
Record Dates: First submitted 2025-09-23; First posted 2025-10-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Breast Cyst; Microcalcification
Keywords: cyst; mass; diagnostic screening; ultrasound; mammography
MeSH Terms: conditions — Breast Neoplasms; Breast Cyst; Calcinosis; Cysts; Arachnodactyly | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Imaging — Ultrasound imaging or ultrasound imaging with light (i.e., photoacoustic imaging)

SUMMARY:
This study aims to investigate recent developments in ultrasound signal processing to determine if these new techniques can enhance the visibility of important features of interest in breast ultrasound images. Ultrasound signals obtained from both standard ultrasound imaging and ultrasound imaging combined with light (also known as photoacoustic imaging) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Female adults (age >18 years) with at least one of the following:
* Macrocalcification(s) detected in x-ray 2D or 3D mammography images
* Macrocalcification(s) located next to cyst (or other identifiable landmark on an ultrasound image)
* A cyst, mass, or finding detected in diagnostic/screening ultrasound or mammography

Exclusion Criteria:

(when performing ultrasound imaging only)

* Children (age < 18 years) are excluded

(when performing ultrasound imaging with light, i.e., optoacoustic imaging)

* Children (age < 18 years) are excluded
* Is pregnant
* Has open sores including insect bites, rash, poison ivy, and chafing on the skin of the ipsilateral breast
* Is experiencing phototoxicity associated with currently taking, or having taken, photosensitizing agents within the previous 72 hours such as sulfonamides, ampicillin, tetracycline
* Is currently undergoing phototherapy
* Has a history of any photosensitive disease (e.g., porphyria, lupus erythematosus) or is undergoing treatment for a photosensitive disease and is experiencing photosensitivity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Johns Hopkins Hospital
Sampling Method: Non-Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2037-01-01 (Estimated); Study Completion 2037-01-01 (Estimated)

PRIMARY OUTCOMES:
Image quality | baseline
  compare advanced beamforming and benchmark against a conventional beamforming technique by measuring and comparing standard image quality metrics
Number of microcalcifications | baseline
Binary visibility of microcalcifications | baseline
  Clinicians (members of study team) will be shown images and record 'yes' if microcalcifications are present and 'no' if not.
Subjective ratings | baseline
  Clinicians (members of study team) will be shown images and asked to provide subjective ratings of the images
Distinction of mass contents: solid vs. fluid | baseline
  After examining the coherence measurements obtained from advanced beamforming techniques, the investigators will determine the ability of this quantitative information to distinguish between solid and fluid-filled masses
Distinction of mass contents: benign vs. malignant | baseline
  After examining the coherence measurements obtained from advanced beamforming techniques, the investigators will determine the ability of this quantitative information to distinguish between solid malignant masses vs. solid benign masses

SECONDARY OUTCOMES:
Number of true positives | baseline
  The number of positive results that are correct
Number of false positives | baseline
  The number of positive results that are incorrect
Number of true negatives | baseline
  The number of negative results that are correct
Number of false negatives | baseline
  The number of negative results that are incorrect

CONTACTS AND LOCATIONS:
Overall Officials: Muyinatu Bell, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No